CLINICAL TRIAL: NCT00699738
Title: Influence of Pregnancy and Post-partum Feeding Method (Breastfeeding Versus Bottlefeeding) on Maternal Hemodynamics (Central and Peripheral) and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008/297
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Healthy women during pregnancy and in the postpartum period
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Healthy women during pregnancy and in the postpartum period, breastfeeding
  Interventions: Behavioral: Breastfeeding
- 2 (Active Comparator): Healthy women during pregnancy and in the postpartum period,bottlefeeding
  Interventions: Behavioral: Bottlefeeding
- 3 (No Intervention): Healthy non-pregnant women

INTERVENTIONS:
Behavioral: Breastfeeding — Breastfeeding
  Arms: 1
Behavioral: Bottlefeeding — Bottlefeeding
  Arms: 2

SUMMARY:
This study will evaluate the physiological and pathophysiological determinants of pregnancy and feeding method on the maternal cardiovascular system. This includes non-invasive measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 40 years old
* Singleton pregnancy
* First pregnancy at the minimum age of 18 years
* In good health, especially no cardiovascular diseases, diabetes or a BMI > 30 kg/m2
* Capable in understanding properly the ICF and the investigators

Exclusion Criteria:

* On chronic medication, especially antihypertensive or antidiabetical drugs
* Multiple pregnancy
* First pregnancy before the age of 18 years old
* Smoking more than 10 cigarettes/day, drinking more than 3 units of alcohol/day or more than 5-6 units of caffeine-containing drinks
* The use of any extralegally drugs
* Not able to have reliable blood pressure or hemodynamic data at screening

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Hemodynamical effects of pregnancy and post-partum feeding method | At approx 8 weeks postpartum.

SECONDARY OUTCOMES:
Effect of the pregnant state and the choice of post-partum feeding method on the parameters of the central and peripheral hemodynamics | At approx 8 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Bortel, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be